CLINICAL TRIAL: NCT05935566
Title: Impact of a History of Tonsillectomy or Adenoidectomy on the Severity of COVID-19 : AMYVID Study
Status: Withdrawn | Type: Observational
Why Stopped: no control patients, so study not launched without comparator
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0052
Record Dates: First submitted 2023-07-05; First posted 2023-07-07 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Tonsillectomy; COVID-19; Adenoidectomy
MeSH Terms: conditions — COVID-19 | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: health questionnaire — Telephone interview with patient to verify medical history, including tonsillectomy and adenoidectomy.

SUMMARY:
Little is known about the impact of tonsillectomy and/or adenoidectomy on the severity and presentation of respiratory infections, let alone COVID-19. Current knowledge of the role of NALT suggests that its absence may be associated with an increased risk of severe disease.

Assessing the impact of tonsillectomy and adenoidectomy on the risk of adverse evolution in COVID-19 would help to better identify patients at risk of adverse evolution, so that they can be rapidly offered appropriate treatment. It would also provide a better understanding of the pathophysiology of this infection.

Primary objective: to determine whether there is a link between a history of tonsillectomy or adenoidectomy and the risk of severe COVID-19.

Primary endpoint: proportion of patients with a history of tonsillectomy or adenoidectomy among those hospitalized for severe COVID-19.

The results of this study will be compared with a data-driven study of Covid patients without severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80
* Hospitalized in SMIT at CHU d'Angers between 01/03/2020 and 30/11/2021 for severe COVID-19 infection (at least 1 severity criterion)

Exclusion Criteria:

Long-term home oxygen therapy prior to COVID-19 infection

* Vaccination against COVID-19 with at least one dose of vaccine received prior to COVID-19 infection Confidential Page 11 of 15
* Inability to ascertain the presence or absence of a history of tonsillectomy or adenoidectomy
* Person objecting to participation in research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at SMIT for severe COVID-19 infection between 01/03/20 and 31/11/21, not previously vaccinated against COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a history of tonsillectomy or adenoidectomy. | immédiat

IPD SHARING:
Plan to Share IPD: No